CLINICAL TRIAL: NCT07232615
Title: A Prospective, Multicenter Clinical Study Comparing Outcomes of Two Trifocal Toric Intraocular Lens
Brief Title: A Planned Study at Multiple Sites is Being Done to Compare the Results of Two Types of Trifocal Toric Intraocular Lenses Used in Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotech Healthcare Holding Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTVCPL-TRITORIC-2019-18
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Presbyopia Correction; Astigmatism; Cataract
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Intervention Model Description: Trifocal Toric Intraocular lens are indicated for primary implantation for visual aphakia secondary to removal of a cataractous lens in adult patients with and without presbyopia who wish to gain near, intermediate and distance vision with decreased dependency on spectacles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Optiflex TRIO (Biotech Europe Meditech Inc. Ltd.) (Experimental): Patients will be implanted with Optiflex TRIO (Biotech Europe Meditech Inc. Ltd.) IOL based on randomization
  Interventions: Device: Optiflex TRIO Intraocular Lens
- AcrySof® IQ PanOptix® (Alcon Laboratories, Inc.) (Active Comparator): Patients will be implanted with AcrySof® IQ PanOptix® (Alcon Laboratories, Inc.) based on randomization
  Interventions: Device: AcrySof® IQ PanOptix®

INTERVENTIONS:
Device: Optiflex TRIO Intraocular Lens — The patients will be implanted with Optiflex TRIO IOL at this arm based on randomization. Trifocal lenses are part of the premium range of refractive-diffractive trifocal IOLs with advanced aspheric optics for excellent visual outcomes. They are single piece, posterior chamber foldable intraocular lenses. The optic is refractive-diffractive trifocal Toric with the anterior surface being aspheric and the posterior surface with a square edge design. The lens is designed to provide all near, distance and intermediate vision and thereby reduce spectacle dependency. Toric version of trifocal intraocular lens is intended to correct astigmatism
  Arms: Optiflex TRIO (Biotech Europe Meditech Inc. Ltd.)
Device: AcrySof® IQ PanOptix® — The patients will be implanted with AcrySof® IQ PanOptix® at this arm based on randomization. Trifocal lenses are part of the premium range of refractive-diffractive trifocal IOLs with advanced aspheric optics for excellent visual outcomes. They are single piece, posterior chamber foldable intraocular lenses. The optic is diffractive trifocal with the anterior surface being aspheric and the posterior surface with a toric component. The lens is designed to provide all near, distance and intermediate vision and thereby reduce spectacle dependency. Toric version of trifocal intraocular lens is intended to correct astigmatism.
  Arms: AcrySof® IQ PanOptix® (Alcon Laboratories, Inc.)

SUMMARY:
To evaluate the clinical outcomes and patient satisfaction of two commercially available trifocal toric intraocular lenses Primary Objective: To compare the distance-corrected intermediate visual acuity between the two trifocal toric intraocular lenses. Secondary Objectives: To assess and compare the safety of two trifocal toric intraocular lenses.

DETAILED DESCRIPTION:
Trifocal lenses are part of the premium range of refractive-diffractive trifocal IOLs with advanced aspheric optics for excellent visual outcomes. They are single piece, posterior chamber foldable intraocular lenses. The optic is refractive-diffractive trifocal with the anterior surface being aspheric and the posterior surface with a square edge design. The lens is designed to provide all near, distance and intermediate vision and thereby reduce spectacle dependency. Toric version of trifocal intraocular lens is intended to correct astigmatism.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patient >21 Years
2. Patient diagnosed with cataract.
3. Patient must have preoperative regular corneal astigmatism between 0.75 to 4.5 D as per corneal topography or keratometry
4. Calculated IOL power is within the range of investigational IOLs.
5. Patient willing to sign inform consent form.
6. Clear intraocular media other than cataract.
7. Female participants of childbearing potential must be willing to ensure that they use effective contraception during the study.

Exclusion Criteria:

1. Previous intraocular or corneal surgery.
2. Traumatic cataract
3. Pregnancy (as stated by patient) or lactation.
4. Concurrent participation in another drug or device investigation.
5. Irregular astigmatism.
6. Patient receiving chlorquine treatment.
7. Subjects with any systemic disease that could increase operative risk or confound the outcome.
8. Active ocular disease in the operative eye other than cataract.
9. Vulnerable subjects as defined in section 12.3.9.
10. Corneal Astigmatism > 4.5 D

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Binocular distance corrected intermediate visual acuity (BCIDVA) | 6 months
  The primary effectiveness endpoint is binocular distance corrected intermediate visual acuity (BCIDVA) at 70 cms at 6 months postoperative, with a target of equivalency between the two IOLs.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (3):
  - Internationale Innovative Ophthalmochirurgie GbR, Düsseldorf, North Rhine-Westphalia
  - Augentagesklinik, Greven, North Rhine-Westphalia
  - Augentagesklinik, Rheine, North Rhine-Westphalia
- India (2):
  - Netradhama Superspeciality Eye Hospital, Bangalore, Karnatak
  - Dr. Agarwal Eye Hospital, Chennai, Tamil Nadu
- Hospital Arruzafa, Córdoba, Córdoba, Spain